CLINICAL TRIAL: NCT01501955
Title: Evaluation of the Safety and Efficiency of the Metaphyseal Hip Prosthesis - Total Hip Arthroplasty
Brief Title: The Metaphyseal Hip Prosthesis - Total Hip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMETEU.CR.EU88 MHP
Record Dates: First submitted 2011-08-26; First posted 2011-12-30 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis of the Hip
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- Stanmore (Active Comparator): 25 patients will have the Stanmore prosthesis
  Interventions: Device: Stanmore
- Metaphyseal Hip Prosthesis (Experimental): 25 patients will have the Metaphyseal Hip Prosthesis (MHP) prosthesis
  Interventions: Device: Metaphyseal Hip Prosthesis

INTERVENTIONS:
Device: Metaphyseal Hip Prosthesis — Metaphyseal Hip Prosthesis (MHP) hip replacement
  Other Names: The Metaphyseal Hip Prosthesis
  Arms: Metaphyseal Hip Prosthesis
Device: Stanmore — Stanmore hip prosthesis
  Other Names: Stanmore hip prosthesis
  Arms: Stanmore

SUMMARY:
The purpose of this study is to analyze stability, safety and efficacy of the Metaphyseal Hip Prosthesis (MHP) compared to the Stanmore hip replacement.

DETAILED DESCRIPTION:
The purpose of this study is to analyze stability, safety and efficacy of the Metaphyseal Hip Prosthesis (MHP) compared to the Stanmore hip replacement at short term (1 year) and long term (10 years).

Bone remodeling will be analyzed at 10 years using DEXA (Dual Energy X-Ray Absorptiometry (bone scan test)) measurements.

This is a single-center prospective study with 25 patients in the study and 25 in the control group in open Randomized Clinical Trial.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for a total hip replacement because of arthritis of the hip
* Patients with a good general condition
* Patients willing and able to participate in the clinical trial with a 10 years follow up and who have signed an inform consent
* Males and females
* Age between 55 and 75
* Absence or little presence of osteoporotic bone (t>-2)
* ASA score 1 and 2

Exclusion Criteria:

* Patient with co morbidities that limit the physical abilities which may negatively influence the scores. Such co morbidities can for example be cardiac insufficiency or chronic respiratory diseases.
* Severe systematic diseases such as rheumatic arthritis and SLE.
* General osteoporosis (t<-2).
* Hormonal conditions such as Paget disease, which reduces the bone density.
* Diseases that can negatively influence the 10 years life expectancy.
* Chronic use of corticosteroids.
* Extreme overweight defined as BMI above 35.
* Active bacterial infection.
* Mental weakness which could negatively influence the postoperative recovery and influence the ability to complete pain scores and other questionnaires.
* ASA score >2.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2023-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stan Bell, MD, Principal Investigator — Bravis Ziekenhuis Roosendaal
Locations (1):
- Bravis Ziekenhuis Roosendaal, Roosendaal, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from all patients eligible for a total hip replacement from either of the investigators at the Bravis Hospital in Roosendaal, between October 2012 and October 2013.
Pre-assignment Details: Pre-operatively a DEXA scan was made to confirm eligibility.
Groups:
- Stanmore: Cemented Stanmore hip stem
- MHP Hip Stem: Cemented MHP (Metaphyseal Hip Prosthesis) hip stem
Period: Overall Study
Arm/Group | Stanmore | MHP Hip Stem
Started | 11 | 9
Surgery | 11 | 9
6 Weeks Postop | 10 (1 patient withdrew on own request) | 9
1 Year Postop | 9 (1 patient terminated due to stem revision) | 7 (2 patients terminated due to stem revision)
2 Years Postop | 9 | 6 (1 patient terminated due to stem revision)
Completed (Primary endpoint at 2 years postop. All active patients will be followed further until 10 years.) | 9 | 6
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 3

BASELINE CHARACTERISTICS:
Population: The population analyzed included all participants with surgery as part of the study. Analysis was performed based on per protocol treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stanmore | MHP Hip Stem | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 9 | 6 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 11 | 9 | 20
Operative Side [Count of Participants; unit: Participants]
  Left | 4 | 3 | 7
  Right | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: RSA Translation X
Description: Stem movement measured with RSA (radiostereometric analysis) along the x-axis in mm. RSA is a technique to accurately measure 3D movement of the prosthesis in the bone. The movement is measured with respect to the situation directly postoperative.
Time Frame: 3 months, 6 months, 1 year and 2 years postoperatively
Population: The population analyzed included all participants with a valid RSA baseline X-ray taken direct postoperatively and with a valid RSA X-ray at the respective time interval. Analysis was performed based on per protocol treatment.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 10 | 7
mm
  3 m postoperatively | 0.05 (0.20) | 0.05 (0.26)
  6 m postoperatively | 0.10 (0.29) | 0.08 (0.35)
  1 y postoperatively: number analyzed (Participants) | 9 | 6
  1 y postoperatively | 0.13 (0.30) | 0.08 (0.41)
  2 y postoperatively: number analyzed (Participants) | 9 | 5
  2 y postoperatively | 0.14 (0.42) | 0.21 (0.60)

2. Primary Outcome: RSA Translation Y
Description: Stem movement along the y-axis in mm. (measured with RSA)
Time Frame: 3 months, 6 months, 1 year and 2 years postoperatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 10 | 7
mm
  3 m postoperatively | -0.25 (0.34) | -0.18 (0.22)
  6 m postoperatively | -0.47 (0.50) | -0.31 (0.28)
  1 y postoperatively: number analyzed (Participants) | 9 | 6
  1 y postoperatively | -0.54 (0.67) | -0.25 (0.24)
  2 y postoperatively: number analyzed (Participants) | 9 | 5
  2 y postoperatively | -0.25 (0.22) | -0.29 (0.43)

3. Primary Outcome: RSA Translation Z
Description: Stem movement along z-axis in mm (measured with RSA)
Time Frame: 3 months, 6 months, 1 year and 2 years postoperatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 10 | 7
mm
  3 m postoperatively | -0.10 (0.36) | -0.08 (0.24)
  6 m postoperatively | -0.23 (0.45) | -0.02 (0.19)
  1 y postoperatively: number analyzed (Participants) | 9 | 6
  1 y postoperatively | -0.19 (0.23) | -0.19 (0.30)
  2 y postoperatively: number analyzed (Participants) | 9 | 5
  2 y postoperatively | -0.25 (0.22) | -0.29 (0.43)

4. Primary Outcome: RSA Rotation X
Description: Stem Rotation around X-axis in degrees (measured with RSA)
Time Frame: 3 months, 6 months, 1 year and 2 years postoperatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 10 | 7
mm
  3 m postoperatively | -0.22 (0.68) | -0.18 (0.13)
  6 m postoperatively | -0.18 (0.74) | -0.23 (1.16)
  1 y postoperatively: number analyzed (Participants) | 9 | 6
  1 y postoperatively | -0.27 (0.48) | -0.44 (0.37)
  2 y postoperatively: number analyzed (Participants) | 9 | 5
  2 y postoperatively | -0.42 (0.92) | -1.18 (0.36)

5. Primary Outcome: RSA Rotation Y
Description: Stem rotation around the y-axis in degrees ( measured with RSA)
Time Frame: 3 months, 6 months, 1 year and 2 years postoperatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 10 | 7
mm
  3 m postoperatively | 0.57 (0.86) | 0.65 (0.59)
  6 m postoperatively | 1.13 (1.36) | 1.22 (1.44)
  1 y postoperatively: number analyzed (Participants) | 9 | 6
  1 y postoperatively | 1.43 (1.29) | 0.52 (0.23)
  2 y postoperatively: number analyzed (Participants) | 10 | 5
  2 y postoperatively | 1.86 (2.00) | 1.50 (0.48)

6. Primary Outcome: RSA Rotation Z
Description: Stem rotation around the z-axis in degrees (measured with RSA)
Time Frame: 3 months, 6 months, 1 year and 2 years postoperatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 10 | 7
mm
  3 m postoperatively | -0.05 (0.28) | -0.26 (0.46)
  6 m postoperatively | -0.01 (0.37) | -0.35 (1.63)
  1 y postoperatively: number analyzed (Participants) | 9 | 6
  1 y postoperatively | -0.11 (0.41) | -0.71 (0.92)
  2 y postoperatively: number analyzed (Participants) | 9 | 5
  2 y postoperatively | -0.08 (0.57) | -1.56 (1.55)

7. Primary Outcome: RSA MTMP
Description: Maximum Total Point Motion (MTPM) measured with RSA. This is a mean for the total migration of the stem.
Time Frame: 3 months, 6 months, 1 year and 2 years postoperatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 10 | 7
mm
  3 m postoperatively | 1.44 (0.79) | 0.81 (0.29)
  6 m postoperatively | 1.75 (1.30) | 1.34 (0.23)
  1 y postoperatively: number analyzed (Participants) | 9 | 6
  1 y postoperatively | 1.76 (1.13) | 1.31 (1.22)
  2 y postoperatively: number analyzed (Participants) | 9 | 5
  2 y postoperatively | 2.48 (1.96) | 3.14 (2.29)

8. Secondary Outcome: Number of Reported Device Related Complications
Description: Safety:
  - Frequency of serious device related complications.
Time Frame: 6 weeks, 3 months, 6 months, 1, 2, 3, 4, 5, 6, 7, 10 years postoperatively
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 11 | 9
participants | 1 | 4

9. Secondary Outcome: Harris Hip Score
Description: Harris Hip Score (HHS), a score to measure health and satisfaction after a hip prosthesis.
  The score has a maximum of 100 points (best possible outcome) covering pain (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 4 points), and range of motion (2 items, 5 points)
Time Frame: pre-operatively, 6 weeks, 3 months, 6 months, 1, 2, 3, 4, 5, 6, 7, and 10 years postoperatively
Population: The population analyzed included all participants with surgery as part of the study. Analysis was performed based on per protocol treatment. Analysis of the Harris Hip Score was performed for all fully completed score forms.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 11 | 9
Scores on a scale
  Pre-operatively: number analyzed (Participants) | 8 | 4
  Pre-operatively | 50.5 (12.0) | 64.0 (10.3)
  6 weeks postoperatively: number analyzed (Participants) | 9 | 6
  6 weeks postoperatively | 90.5 (9.6) | 83.8 (10.3)
  3 months postoperatively: number analyzed (Participants) | 9 | 7
  3 months postoperatively | 91.3 (7.6) | 83.8 (12.2)
  6 months postoperatively: number analyzed (Participants) | 9 | 6
  6 months postoperatively | 94.8 (6.4) | 82.2 (18.8)
  1 year postoperatively: number analyzed (Participants) | 8 | 8
  1 year postoperatively | 95.6 (5.7) | 80.6 (20.7)
  2 years postoperatively: number analyzed (Participants) | 6 | 4
  2 years postoperatively | 94.9 (1.8) | 81.0 (15.6)
  3 years postoperatively: number analyzed (Participants) | 8 | 4
  3 years postoperatively | 94.9 (1.8) | 95.9 (0.0)
  4 years postoperatively: number analyzed (Participants) | 7 | 3
  4 years postoperatively | 92.0 (8.6) | 85.2 (18.5)
  5 years postoperatively: number analyzed (Participants) | 3 | 3
  5 years postoperatively | 94.6 (2.3) | 91.6 (5.9)
  6 years postoperatively: number analyzed (Participants) | 3 | 2
  6 years postoperatively | 93.6 (4.0) | 77.4 (3.5)
  7 years postoperatively: number analyzed (Participants) | 3 | 0
  7 years postoperatively | 92.7 (2.9) |
  10 years postoperatively: number analyzed (Participants) | 3 | 2
  10 years postoperatively | 87.5 (14.5) | 96.0 (0.1)

10. Secondary Outcome: DEXA
Description: Efficacy: Bone density measured using the average DEXA score in each zone. For the long Stanmore the 7 Gruen zones were defined. For the short MHP stem an adjusted model with only 5 zones was used. The scan at 6 weeks is used as the baseline measurement to analyze if the bone density changes in the following years. At 1 year and 2 year follow up, percentual change is presented for both groups with respect to the 6 weeks DEXA score
Time Frame: 1 and 2 years postoperative
Population: The population analyzed included all participants with surgery as part of the study. Analysis was performed based on per protocol treatment. Percentage of change was calculated for all participants that have paired results available (6 week and 1 year or 6 week and 2 year). For MHP stem only 5 Gruen Zones were defined, so no information available for zone 6 and 7.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 8 | 6
percentage of change
  Zone 1 - 1 year PO | 10.8 (51.4) | 6.8 (54.7)
  Zone 1 - 2 year PO: number analyzed (Participants) | 8 | 5
  Zone 1 - 2 year PO | -4.8 (11.4) | -8.1 (34.1)
  Zone 2 - 1 year PO | -8.1 (17.7) | -17.7 (26.7)
  Zone 2 - 2 year PO: number analyzed (Participants) | 8 | 5
  Zone 2 - 2 year PO | -2.0 (4.5) | -6.3 (32.3)
  Zone 3 - 1 year PO | -3.5 (7.2) | -7.4 (15.4)
  Zone 3 - 2 year PO: number analyzed (Participants) | 8 | 5
  Zone 3 - 2 year PO | -3.5 (7.2) | -9.9 (14.3)
  Zone 4 - 1 year PO | 4.3 (5.0) | -0.8 (35.2)
  Zone 4 - 2 year PO: number analyzed (Participants) | 8 | 5
  Zone 4 - 2 year PO | 0.3 (13.2) | -4.5 (37.9)
  Zone 5 - 1 year PO | 4.4 (6.1) | -21.3 (28.7)
  Zone 5 - 2 year PO: number analyzed (Participants) | 8 | 5
  Zone 5 - 2 year PO | 6.5 (10.6) | -19.1 (35.9)
  Zone 6 - 1 year PO: number analyzed (Participants) | 8 | 0
  Zone 6 - 1 year PO | 2.0 (5.9) |
  Zone 6 - 2 year PO: number analyzed (Participants) | 8 | 0
  Zone 6 - 2 year PO | -1.7 (9.4) |
  Zone 7 - 1 year PO: number analyzed (Participants) | 8 | 0
  Zone 7 - 1 year PO | 8.4 (27.7) |
  Zone 7 - 2 year PO: number analyzed (Participants) | 8 | 0
  Zone 7 - 2 year PO | 8.4 (27.7) |

11. Secondary Outcome: HOOS-Pain Subscale
Description: HOOS (Hip disability and Osteoarthritis Outcome Score) consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and hip related Quality of life (QOL). The last week is taken into consideration when answering the questions. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Time Frame: pre-operatively, 6 weeks, 3 months, 6 months, 1, 2, 3, 4, 5, 6, 7, and 10 years postoperatively
Population: The population analyzed included all participants with surgery as part of the study. Analysis was performed based on per protocol treatment. Analysis of the HOOS Score was performed for all valid completed score forms.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 10 | 9
units on a scale
  Pre-operatively | 44.4 (19.7) | 51.7 (27.8)
  6 weeks postoperatively: number analyzed (Participants) | 8 | 8
  6 weeks postoperatively | 84.2 (11.3) | 74.7 (23.3)
  3 months postoperatively: number analyzed (Participants) | 7 | 7
  3 months postoperatively | 78.6 (15.1) | 76.1 (21.8)
  6 months postoperatively: number analyzed (Participants) | 9 | 7
  6 months postoperatively | 87.2 (21.3) | 73.9 (24.7)
  1 year postoperatively: number analyzed (Participants) | 9 | 7
  1 year postoperatively | 95.8 (8.0) | 78.2 (29.5)
  2 years postoperatively: number analyzed (Participants) | 9 | 6
  2 years postoperatively | 84.8 (18.2) | 84.7 (27.6)
  3 years postoperatively: number analyzed (Participants) | 9 | 3
  3 years postoperatively | 86.1 (16.8) | 100.0 (0.0)
  4 years postoperatively: number analyzed (Participants) | 9 | 4
  4 years postoperatively | 88.5 (16.6) | 87.5 (25.0)
  5 years postoperatively: number analyzed (Participants) | 9 | 3
  5 years postoperatively | 87.8 (16.7) | 98.3 (2.9)
  6 years postoperatively: number analyzed (Participants) | 5 | 4
  6 years postoperatively | 80.0 (26.3) | 89.4 (21.3)
  7 years postoperatively: number analyzed (Participants) | 7 | 4
  7 years postoperatively | 91.1 (7.5) | 91.3 (17.5)
  10 years postoperatively: number analyzed (Participants) | 5 | 3
  10 years postoperatively | 86.5 (17.6) | 100.0 (0.0)

12. Secondary Outcome: HOOS-Symptom Subscale
Description: HOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and hip related Quality of life (QOL). The last week is taken into consideration when answering the questions. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Time Frame: pre-operatively, 6 weeks, 3 months, 6 months, 1, 2, 3, 4, 5, 6, 7, and 10 years postoperatively
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 11 | 9
units on a scale
  Pre-operatively | 39.5 (16.2) | 57.2 (25.0)
  6 weeks postoperatively: number analyzed (Participants) | 9 | 8
  6 weeks postoperatively | 74.4 (14.4) | 63.1 (22.7)
  3 months postoperatively: number analyzed (Participants) | 8 | 7
  3 months postoperatively | 68.8 (18.5) | 70.7 (19.0)
  6 months postoperatively: number analyzed (Participants) | 10 | 7
  6 months postoperatively | 76.0 (22.8) | 75.0 (16.8)
  1 year postoperatively: number analyzed (Participants) | 9 | 7
  1 year postoperatively | 89.0 (11.0) | 70.7 (31.5)
  2 years postoperatively: number analyzed (Participants) | 9 | 6
  2 years postoperatively | 85.0 (11.5) | 86.7 (14.7)
  3 years postoperatively: number analyzed (Participants) | 9 | 3
  3 years postoperatively | 84.7 (16.4) | 96.7 (5.8)
  4 years postoperatively: number analyzed (Participants) | 9 | 4
  4 years postoperatively | 85.0 (14.4) | 82.5 (25.3)
  5 years postoperatively: number analyzed (Participants) | 9 | 3
  5 years postoperatively | 90.8 (9.4) | 96.7 (5.8)
  7 years postoperatively: number analyzed (Participants) | 7 | 4
  7 years postoperatively | 90.7 (6.7) | 83.8 (20.2)
  10 years postoperatively: number analyzed (Participants) | 5 | 3
  10 years postoperatively | 82.0 (15.2) | 81.7 (16.1)

13. Secondary Outcome: HOOS-ADL Subscale
Description: as for outcome 12
Time Frame: pre-operatively, 6 weeks, 3 months, 6 months, 1, 2, 3, 4, 5, 6, 7, and 10 years postoperatively
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 11 | 9
units on a scale
  Pre-operatively | 46.6 (17.8) | 52.4 (27.7)
  6 weeks postoperatively: number analyzed (Participants) | 8 | 8
  6 weeks postoperatively | 76.4 (14.5) | 77.77 (28.0)
  3 months postoperatively: number analyzed (Participants) | 8 | 7
  3 months postoperatively | 81.4 (15.6) | 78.0 (23.5)
  6 months postoperatively: number analyzed (Participants) | 10 | 7
  6 months postoperatively | 84.5 (16.7) | 75.6 (23.5)
  1 year postoperatively: number analyzed (Participants) | 9 | 7
  1 year postoperatively | 92.2 (8.5) | 73.7 (31.8)
  2 years postoperatively: number analyzed (Participants) | 9 | 6
  2 years postoperatively | 86.2 (14.0) | 90.9 (17.5)
  3 years postoperatively: number analyzed (Participants) | 9 | 3
  3 years postoperatively | 87.8 (15.1) | 100.0 (0.0)
  4 years postoperatively: number analyzed (Participants) | 9 | 4
  4 years postoperatively | 87.7 (15.4) | 90.4 (19.2)
  5 years postoperatively: number analyzed (Participants) | 8 | 3
  5 years postoperatively | 88.4 (17.2) | 99.0 (1.7)
  6 years postoperatively: number analyzed (Participants) | 5 | 4
  6 years postoperatively | 82.8 (23.9) | 91.5 (16.9)
  7 years postoperatively: number analyzed (Participants) | 7 | 4
  7 years postoperatively | 91.0 (8.8) | 90.1 (19.9)
  10 years postoperatively: number analyzed (Participants) | 5 | 3
  10 years postoperatively | 81.6 (21.6) | 95.8 (7.2)

14. Secondary Outcome: HOOS-Sport Subscale
Description: as for outcome 12
Time Frame: pre-operatively, 6 weeks, 3 months, 6 months, 1, 2, 3, 4, 5, 6, 7, and 10 years postoperatively
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 11 | 9
units on a scale
  Pre-operatively: number analyzed (Participants) | 11 | 8
  Pre-operatively | 27.3 (17.5) | 26.6 (21.8)
  6 weeks postoperatively: number analyzed (Participants) | 7 | 6
  6 weeks postoperatively | 56.3 (25.3) | 40.3 (30.7)
  3 months postoperatively: number analyzed (Participants) | 8 | 6
  3 months postoperatively | 59.4 (29.3) | 50.0 (33.8)
  6 months postoperatively: number analyzed (Participants) | 10 | 6
  6 months postoperatively | 63.1 (28.8) | 48.3 (37.0)
  1 year postoperatively: number analyzed (Participants) | 8 | 6
  1 year postoperatively | 75.8 (25.3) | 41.7 (30.8)
  2 years postoperatively: number analyzed (Participants) | 9 | 5
  2 years postoperatively | 68.8 (21.0) | 80.0 (30.4)
  3 years postoperatively: number analyzed (Participants) | 8 | 2
  3 years postoperatively | 73.4 (27.4) | 100.0 (0.0)
  4 years postoperatively: number analyzed (Participants) | 8 | 3
  4 years postoperatively | 71.9 (23.9) | 70.8 (50.5)
  5 years postoperatively: number analyzed (Participants) | 8 | 1
  5 years postoperatively | 71.9 (23.9) | 100.0
  6 years postoperatively: number analyzed (Participants) | 6 | 2
  6 years postoperatively | 67.7 (41.9) | 62.5 (53.0)
  7 years postoperatively: number analyzed (Participants) | 7 | 2
  7 years postoperatively | 69.9 (19.0) | 71.9 (39.8)
  10 years postoperatively: number analyzed (Participants) | 5 | 1
  10 years postoperatively | 59.2 (28.6) | 100.0

15. Secondary Outcome: HOOS-QoL Subscale
Description: as for outcome 12
Time Frame: pre-operatively, 6 weeks, 3 months, 6 months, 1,2, 3, 4, 5, 6, 7, and 10 years postoperatively
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 11 | 9
units on a scale
  Pre-operatively | 34.8 (14.6) | 34.5 (26.5)
  6 weeks postoperatively: number analyzed (Participants) | 8 | 8
  6 weeks postoperatively | 60.2 (15.7) | 60.1 (31.0)
  3 months postoperatively: number analyzed (Participants) | 8 | 7
  3 months postoperatively | 59.4 (23.4) | 62.5 (40.8)
  6 months postoperatively: number analyzed (Participants) | 10 | 7
  6 months postoperatively | 74.6 (22.8) | 59.8 (38.7)
  1 year postoperatively: number analyzed (Participants) | 8 | 7
  1 year postoperatively | 89.8 (16.0) | 68.8 (40.3)
  2 years postoperatively: number analyzed (Participants) | 9 | 6
  2 years postoperatively | 81.9 (19.6) | 81.9 (40.3)
  3 years postoperatively: number analyzed (Participants) | 9 | 3
  3 years postoperatively | 80.6 (28.7) | 100.0 (0.0)
  4 years postoperatively: number analyzed (Participants) | 9 | 4
  4 years postoperatively | 84.0 (18.0) | 75.0 (50.0)
  5 years postoperatively: number analyzed (Participants) | 9 | 2
  5 years postoperatively | 86.8 (18.6) | 100.0 (0.0)
  6 years postoperatively: number analyzed (Participants) | 6 | 4
  6 years postoperatively | 100.0 (0.0) | 78.1 (43.8)
  7 years postoperatively: number analyzed (Participants) | 7 | 4
  7 years postoperatively | 92.9 (14.2) | 75.0 (50.0)
  10 years postoperatively: number analyzed (Participants) | 5 | 3
  10 years postoperatively | 88.3 (14.3) | 93.8 (10.8)

16. Secondary Outcome: SF-12 Physical Summary Score
Description: 12-Item Short-Form Health Survey (SF-12) presented in Physical (PS) and Mental summary (MS) scores (range 0-100).
  A zero score indicates the lowest level of health and 100 indicates the highest level of health.
Time Frame: pre-operatively, 6 weeks, 3 months, 6 months, 1, 2, 3, 4, 5, 6, 7, and 10 years postoperatively
Population: The population analyzed included all participants with surgery as part of the study. Analysis was performed based on per protocol treatment. Analysis of the SF-12 Score was performed for all fully completed score forms.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 11 | 9
units on a scale
  Pre-operatively | 34.7 (6.4) | 37.3 (8.7)
  6 weeks postoperatively: number analyzed (Participants) | 10 | 8
  6 weeks postoperatively | 44.2 (7.3) | 41.3 (9.0)
  3 months postoperatively: number analyzed (Participants) | 8 | 7
  3 months postoperatively | 42.4 (7.3) | 43.0 (12.5)
  6 months postoperatively: number analyzed (Participants) | 10 | 7
  6 months postoperatively | 46.5 (8.0) | 42.7 (11.0)
  1 year postoperatively: number analyzed (Participants) | 9 | 7
  1 year postoperatively | 51.6 (4.5) | 48.7 (8.2)
  2 years postoperatively: number analyzed (Participants) | 9 | 6
  2 years postoperatively | 48.4 (8.9) | 54.4 (3.1)
  3 years postoperatively: number analyzed (Participants) | 9 | 3
  3 years postoperatively | 47.3 (9.6) | 53.3 (3.5)
  4 years postoperatively: number analyzed (Participants) | 9 | 4
  4 years postoperatively | 45.9 (6.7) | 50.6 (7.5)
  5 years postoperatively: number analyzed (Participants) | 9 | 4
  5 years postoperatively | 49.2 (7.7) | 53.6 (3.1)
  6 years postoperatively: number analyzed (Participants) | 6 | 4
  6 years postoperatively | 41.2 (7.7) | 49.1 (8.8)
  7 years postoperatively: number analyzed (Participants) | 7 | 4
  7 years postoperatively | 48.1 (6.4) | 46.3 (9.7)
  10 years postoperatively: number analyzed (Participants) | 5 | 3
  10 years postoperatively | 48.4 (7.5) | 48.4 (5.2)

17. Secondary Outcome: SF-12 Mental Summary Score
Description: SF-12 Score presented in Physical and Mental summary scores (range 0-100). A zero score indicates the lowest level of health and 100 indicates the highest level of health.
Time Frame: pre-operatively, 6 weeks, 3 months, 6 months, 1, 2, 3, 4, 5, 6, 7, and 10 years postoperatively
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stanmore | MHP Hip Stem
Number analyzed (Participants) | 11 | 9
units on a scale
  Pre-operatively | 53.7 (7.6) | 53.5 (12.4)
  6 weeks postoperatively: number analyzed (Participants) | 10 | 8
  6 weeks postoperatively | 56.9 (3.7) | 50.8 (11.6)
  3 months postoperatively: number analyzed (Participants) | 8 | 7
  3 months postoperatively | 59.7 (2.8) | 53.1 (9.4)
  6 months postoperatively: number analyzed (Participants) | 10 | 7
  6 months postoperatively | 59.0 (3.5) | 49.1 (9.4)
  1 year postoperatively: number analyzed (Participants) | 9 | 7
  1 year postoperatively | 56.5 (8.1) | 50.1 (11.7)
  2 years postoperatively: number analyzed (Participants) | 9 | 6
  2 years postoperatively | 57.5 (6.3) | 55.4 (6.8)
  3 years postoperatively: number analyzed (Participants) | 9 | 3
  3 years postoperatively | 58.8 (7.9) | 59.8 (1.6)
  4 years postoperatively: number analyzed (Participants) | 9 | 4
  4 years postoperatively | 60.5 (3.0) | 57.0 (7.1)
  5 years postoperatively: number analyzed (Participants) | 9 | 4
  5 years postoperatively | 52.7 (7.6) | 57.7 (4.0)
  6 years postoperatively: number analyzed (Participants) | 6 | 4
  6 years postoperatively | 54.1 (10.3) | 57.2 (5.6)
  7 years postoperatively: number analyzed (Participants) | 7 | 4
  7 years postoperatively | 56.8 (2.9) | 52.4 (10.1)
  10 years postoperatively: number analyzed (Participants) | 5 | 3
  10 years postoperatively | 53.6 (10.8) | 58.9 (0.8)

ADVERSE EVENTS:
Time Frame: SAE´s collected up to 10 years post/operatively
Description: The occurrence of adverse events was assessed at each follow up visit.
Arm/Group | Stanmore | MHP Hip Stem
All-Cause Mortality (participants affected / at risk) | 1/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 2/11 | 7/9
Other Adverse Events (participants affected / at risk) | 2/11 | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stanmore (N=11) | MHP Hip Stem (N=9)
Stem revision (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Cardiac Disorder (Cardiac disorders) | 1 (1) | 1 (1) — ST depression and Myocard Infarction
Cup revision (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stanmore (N=11) | MHP Hip Stem (N=9)
Cortical Erosion/Osteolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in groin During Weigth Bearing (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Superficial Infection Wound (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The enrollment was terminated early leading to a small number of patients available for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT01501955/Prot_SAP_000.pdf